CLINICAL TRIAL: NCT06503523
Title: Investigation of the Neurophysiological and Psychological Aspects of Itch
Brief Title: The Effects of Performing a Motor Imagery Task on Cortical Excitability During Acute Experimental Muscle Pain and Acute Itch
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20240004 2nd subproject
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Itch; Pain
MeSH Terms: conditions — Pruritus; Pain | interventions — Saline Solution, Hypertonic; Histamine; Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: we apply one of three experimental methods in your hand: either an injection of salt water (7% NaCl) or we apply small needles from the plant mucuna pruriens or histamine (1%)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental:Healthy volunteers (Experimental)
  Interventions: Other: Hypertonic Saline; Other: Histamine; Other: Cowhage; Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Other: Hypertonic Saline — A bolus injection of hypertonic saline (7% NaCl) will be administered to the FDI muscle using a 1 mL syringe with a disposable needle (27G), and the volume of the bolus will be 0.1 mL
Other: Histamine — A small drop of histamine dihydrochloride will be applied to a previously determined area on the volar forearm, followed by a prick through the drop
Other: Cowhage — This insertion is conducted by forceps using a stereomicroscope, and 30-35 spicules are gently rubbed into a 1 cm diameter skin area.
Device: Transcranial magnetic stimulation (TMS) — Transcranial magnetic stimulation (TMS) will be used to evoke motor-evoked potentials (MEPs) in the muscle of interest and cortical responses (TMSevoked potentials - TEPs) in the motor cortex with a figure-eight-shaped cone coil.

SUMMARY:
The aim of this project is to determine the effects of performing a motor imagery task on cortical excitability during acute experimental muscle pain (induced by hypertonic saline), acute histaminergic itch (induced by histamine), and non-histaminergic itch stimulation (triggered by Cowhage). We hypothesize that motor imagery will counteract the alterations in cortical excitability observed during experimental muscle pain and both itch models.

DETAILED DESCRIPTION:
Itch and pain share many similarities and dissimilarities in terms of the mechanisms and molecules involved. Many studies have been conducted to explain all the neurophysiological aspects involved in the pain process, and cortical adaptations have been provoked in healthy individuals using experimental pain models. Unfortunately, all these aspects still need to be clarified regarding itch. Has been previously demonstrated that motor imagery can counteracted the pain-induced decrease in corticospinal excitability observed during acute pain, and it has also been proposed as a potential intervention for individuals with pain to restore maladaptive neuroplasticity. However, whether motor imagery can similarly counteract the itch-induced cortical changes remains unclear. Therefore, the aim of this project is to investigate whether motor imagery would counteract the reduction in cortical excitability during acute itch, similar to the effects observed in the context of acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g. neuropathy), immunological (e.g. asthma, immune deficiencies, arthritis), musculoskeletal (e.g. muscular pain in the upper extremities,), cardiac disorder (e.g., heart stroke), or psychiatric diagnoses (e.g. depression) that may affect the results
* Current use of medications that may affect the trial, such as antihistamines, antipsychotics, and painkillers, as well as systemic or topical steroids
* Skin diseases (e.g., atopic dermatitis, pruritus nodularis, eczema, psoriasis)
* Moles, scars, or tattoos in the area to be treated or tested.
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain
* Unable to pass the "Transcranial Magnetic Stimulation Adult Safety Screen" (subproject 1 and 2)
* Contraindications to transcranial magnetic stimulation (TMS) application (history of epilepsy, metal implants in head or jaw, etc.)
* Presence of implanted hearing aids or metal implants on the face, including permanent makeup or tattoos
* Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scales (NRS) | 1 minute after every itch/pain induction
  NRS are essentially VAS but have tick marks spaced every centimeter so as to create 11-point scale (from 0 to 10).
  Subject can use these tick marks as a guide when they mark their severity on the scale.
Measuring cortical excitability (TEPs) | Baseline
  Transcranial magnetic stimulation (TMS) with a figure-eight-shaped cone coil will be used to evoke cortical responses in the motor cortex. The resulting TMS-evoked potentials (TEPs) will be collected using an electroencephalogram (EEG). This assessment will last for 7 minutes before inducing itch or pain.
Measuring cortical excitability (TEPs) | During Itch/pain stimulation for 10 minutes
  Transcranial magnetic stimulation (TMS) with a figure-eight-shaped cone coil will be used to evoke cortical responses in the motor cortex. The resulting TMS-evoked potentials (TEPs) will be collected using an electroencephalogram (EEG). This assessment will last for 7 minutes during itch or pain. The pain or itch sensation will last 10 minutes.
Measuring cortical excitability (TEPs) | During motor imagery task for 7 minutes
  Transcranial magnetic stimulation (TMS) with a figure-eight-shaped cone coil will be used to evoke cortical responses in the motor cortex. The resulting TMS-evoked potentials (TEPs) will be collected using an electroencephalogram (EEG). This assessment will last for 7 minutes during motor imagery task.
Measuring cortical excitability (TEPs) | Post induction of itch or pain
  Transcranial magnetic stimulation (TMS) with a figure-eight-shaped cone coil will be used to evoke cortical responses in the motor cortex. The resulting TMS-evoked potentials (TEPs) will be collected using an electroencephalogram (EEG). Similar to the baseline, this assessment will last for 7 minutes after itch or pain.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS). | Baseline
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Itch Catastrophizing Scale (ICS). | Baseline
  The ICS assesses negative and exaggerated coping concerning anticipated or experienced itchy stimuli. Thirteen items have to be answered on a 5-point Likert-type scale.
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline
  The RST-PQ contains the following subscales: the Fight-Flight-Freeze System (FFFS, 10 items), which represents a defensive factor related to active avoidance of adverse stimuli; the Behavioral Inhibition System (BIS, 23 items), which represents a defensive factor related to anxiety and passive avoidance of adverse stimuli; and the Behavioral Approach System (BAS, 32 items), which reflects reward interest, goal-drive persistence, reward reactivity, and impulsivity. In total, 65 items have to be answered on a 4-point Likert-type scale
The Pittsburg Sleep Quality Index (PSQI) | Baseline
  The PSQI consists of 19 items generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The seven component scores can be summarized in a global score ranging from zero to 21 with higher scores reflecting a worse overall quality of sleep
Depression, Anxiety, Stress Scale (DASS-21) | Baseline
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much".
Learned Helplessness Scale (LHS) | Baseline
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale ranging from strongly agree (1) to strongly disagree (4).
Positive And Negative Affect Schedule (PANAS) | Baseline
  PANAS measures positive and negative affect dimensions. Twenty words are associated with the subject's current feelings and have to be rated on a 5-points Likert-type scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark